CLINICAL TRIAL: NCT07312448
Title: Single-Center Retrospective Comparative Analysis Of Modified Vs. Classical Nuss Technique In The Surgical Correction Of Pectus Excavatum "
Brief Title: Comparative Analysis Of Modified Vs. Classical Nuss Technique In The Surgical Correction Of Pectus Excavatum "
Acronym: PE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9450
Record Dates: First submitted 2025-12-09; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pectus Excavatum
Keywords: Pectus Excavatum; Nuss techniques; Modified Nuss Technique
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although the NUSS technique has become the standard minimally invasive procedure for correcting this deformity, there is a lack of comparative data between the classic and modified NUSS techniques. This research aims to fill this gap by comparing these two methods in terms of various outcomes, such as operative time, postoperative pain control, length of stay in the intensive care unit, and overall cosmetic results.

This study addresses the need to optimize surgical techniques to improve patient outcomes. By evaluating these two approaches, the research seeks to provide insights that could lead to better management strategies for patients with pectus excavatum, potentially influencing future clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 11 to 18 years.
* Patients who underwent surgery between 2010 and 2024 using either the classic or modified Nuss technique. - Patient with a Haller index of 2.25 or higher.

Exclusion Criteria:

* Patients with a Haller score below 2.25.
* Patients who have undergone surgery using alternative techniques such as Ravitch or modified Ravitch.
* Patients under 11 years of age or over 19 years of age.

Ages: 11 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients aged 11 to 18 years underwent surgery between 2010 and 2024 using either the classic or modified Nuss technique. - Patient with a Haller index of 2.25 or higher.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Operating time (in minutes) | Operating time (in minutes)
  Comparaison Of Modified Vs. Classical Nuss Technique In The Surgical Correction Of Pectus Excavatum in terms of operating time criterion (in minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Pédiatrique - Réanimation - CHU de Strasbourg - France, Strasbourg, France